CLINICAL TRIAL: NCT00705406
Title: A Phase II, Multicenter, Randomized, Placebo -Controlled, Study To Evaluate The Efficacy and Safety Of Intramuscular Peramivir 600 mg In Subjects With Uncomplicated Acute Influenza
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCX1812-212; HHS 0100200700032C (Other Grant/Funding Number: HHS-BARDA)
Record Dates: First submitted 2008-06-24; First posted 2008-06-26 (Estimated); Results first posted 2015-02-16 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Acute, Uncomplicated Human Influenza
MeSH Terms: interventions — peramivir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peramivir 600 mg (Experimental): 600 mg peramivir administered as bilateral 2-mL intramuscular injection.
  Interventions: Drug: Peramivir
- Placebo (Placebo Comparator): Placebo (buffered diluent) administered as bilateral 2-mL intramuscular injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Peramivir — 600 mg peramivir administered as bilateral 2-mL intramuscular injection
  Arms: Peramivir 600 mg
Drug: Placebo — Placebo (buffered diluent) administered as bilateral 2-mL intramuscular injection.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether peramivir is safe and effective in the treatment of uncomplicated seasonal influenza.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female subjects age ≥18 years.
* A positive Influenza A or B Rapid Antigen Test (RAT) performed with a commercially available test kit on an adequate anterior nasal specimen, in accordance with the manufacturer's instructions. A negative initial RAT should be repeated within one hour.
* Presence of fever at time of screening of ≥38.0 ºC (≥100.4 ºF) taken orally, or ≥38.5 ºC (≥101.2 ºF) taken rectally. A subject self-report of a history of fever or feverishness within the 24 hours prior to screening will also qualify for enrollment in the absence of documented fever at the time of screening.
* Presence of at least one respiratory symptom (cough, sore throat, or nasal symptoms) of at least moderate severity.
* Presence of at least one constitutional symptom (myalgia [aches and pains], headache, feverishness, or fatigue) of at least moderate severity.
* Onset of symptoms no more than 36 hours before presentation for screening.
* Written informed consent.

Exclusion Criteria:

* Women who are pregnant or breast-feeding.
* Presence of clinically significant signs of acute respiratory distress
* History of severe chronic obstructive pulmonary disease (COPD) or severe persistent asthma.
* History of heart failure or angina requiring daily pharmacotherapy with symptoms consistent with New York Heart Association Class III or IV functional status within the past 12 months.
* Screening ECG which suggests acute ischemia or presence of medically significant dysrhythmia.
* History of chronic renal impairment requiring hemodialysis and/or known or suspected to have moderate or severe renal impairment (actual or estimated creatinine clearance <50 mL/min).
* Clinical evidence of worsening of any chronic medical condition (temporally associated with the onset of symptoms of influenza) which, in the investigator's opinion, indicates that such finding(s) could represent complications of influenza.
* Current clinical evidence, including clinical signs and/or symptoms consistent with otitis, bronchitis, sinusitis and/or pneumonia, or active bacterial infection at any body site that requires therapy with oral or systemic antibiotics.
* Presence of immunocompromised status due to chronic illness, previous organ transplant, or use of immunosuppressive medical therapy which would include oral or systemic treatment with > 10 mg prednisone or equivalent on a daily basis within 30 days of screening.
* Currently receiving treatment for viral hepatitis B or viral hepatitis C.
* Presence of known HIV infection with a CD4 count <350 cell/mm3.
* Current therapy with oral warfarin or other systemic anticoagulant.
* Receipt of any doses of rimantadine, amantadine, zanamivir, or oseltamivir in the 7 days prior to screening.
* Immunized against influenza with live attenuated virus vaccine (FluMist®) in the previous 21 days.
* Immunized against influenza with inactivated virus vaccine within the previous 14 days.
* Receipt of any intramuscular injection with the previous 7 days.
* History of alcohol abuse or drug addiction within 1 year prior to admission in the study.
* Participation in a previous study of intramuscular or intravenous peramivir or previous participation in this study.
* Participation in a study of any investigational drug or device within the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2008-07; Primary Completion 2009-04 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (122):
- United States (66):
  - West Alabama Research, Inc., Birmingham, Alabama
  - Greystone Medical Research, LLC, Birmingham, Alabama
  - NextCare Institute for Clinical Research, Phoenix, Arizona
  - Clopton Clinic, Jonesboro, Arkansas
  - NEA Clinic, Jonesboro, Arkansas
  - North Central Arkansas Medical Associates, Mountain Home, Arkansas
  - Impact Clinical Trials, Beverly Hills, California
  - Medcenter, Carmichael, California
  - Center for Clinical Trials, LLC, Paramount, California
  - Coastal Medical Research Group, Inc., San Luis Obispo, California
  - Alpine Research Center, Boulder, Colorado
  - 1st Allergy and Clinical Research Center, Centennial, Colorado
  - Clinical Research of South Florida, Coral Gables, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - University Clinical Research, Inc., Pembroke Pines, Florida
  - DMI Research, Inc., Pinellas Park, Florida
  - Wilker/Powers Center for Clinical Studies, d/b/a ProHealth Clinical Studies, Saint Cloud, Florida
  - Southeast Regional Research Group, Columbus, Georgia
  - Southeast Regional Research Group, Savannah, Georgia
  - The Kaufmann Clinic, Inc., Woodstock, Georgia
  - Idaho Falls Infectious Diseases, Idaho Falls, Idaho
  - Dr. Arthur Davida, Bloomingdale, Illinois
  - Investigators Research Group, LLC, Indianapolis, Indiana
  - Medical Associates Clinic, Dubuque, Iowa
  - Heart of America Research, Shawnee, Kansas
  - Kentucky Lung Clinic, Hazard, Kentucky
  - Gulf Coast Research, LLC, Baton Rouge, Louisiana
  - Acadia Clinical Research, Bangor, Maine
  - Clarksburg Medical Center, Clarksburg, Maryland
  - Miray Medical Center, Brockton, Massachusetts
  - Detroit Receiving Hospital, UHC 6G, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - KMED Research, Saint Claire Shores, Michigan
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - Bozeman Urgent Care Center, Bozeman, Montana
  - Mercury Street Medical Group, PLLC, Butte, Montana
  - Prairie Fields Family Medicine, P.C., Fremont, Nebraska
  - Impact Clinical Trials, Las Vegas, Las Vegas, Nevada
  - United Medical Associates, Johnson City, New York
  - Twelve Corners Internal Medicine, Rochester, New York
  - Bland Clinic, Greensboro, North Carolina
  - Community Medical Associates, LLC, Canfield, Ohio
  - Advanced Health Care Services, Inc, Thornville, Ohio
  - Urgent Care of Green County, PLLC, Owasso, Oklahoma
  - Integrated Medical Research, PC, Ashland, Oregon
  - Pivotal Clinical Research, LLC, Souderton, Pennsylvania
  - New England Center for Clinical Research, Inc., Cranston, Rhode Island
  - Notheast Clinical Research, Cumberland, Rhode Island
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Omega Medical Research, Warwick, Rhode Island
  - Hillcrest Clinical Research, LLC, Simpsonville, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - Holston Medical Group, Bristol, Tennessee
  - DiscoveResearch, Inc., Bryan, Texas
  - Corpus Christi Family Wellness Center, Research Division, Corpus Christi, Texas
  - Allergy/Immunology Research Center of North Texas, Dallas, Texas
  - Towngate Plaza Medical Center, Garland, Texas
  - West Houston Clinical Research, Houston, Texas
  - Texas Medical Research Associates, LLC, San Antonio, Texas
  - Martin Diagnostic Clinic, Tomball, Texas
  - J. Lewis Research, Inc., FirstMed, Salt Lake City, Utah
  - J. Lewis Research, Inc./Foothill Family Clinic South, Salt Lake City, Utah
  - J. Lewis Research, Inc./FirstMed East, Salt Lake City, Utah
  - Northwest Clinical Research Center, Bellevue, Washington
  - Dean Medical Center, Oregon, Wisconsin
- Australia (15):
  - Pacific Medical Centre Blacktown, Blacktown, New South Wales
  - East Sydney Doctors, Darlinghurst, New South Wales
  - Symbion Pathology, Hurtsville, New South Wales
  - Peninsula Medical Centre, Umina, New South Wales
  - Rivercity Private Hospital Specialist, Auchenflower, Queensland
  - Caboolture Clinical Research Centre, Caboolture, Queensland
  - Peninsula Specialist Centre, Kpparing, Queensland
  - Health Services -University of Melbourne, Carlton, Victoria
  - Athelstone Medical Clinic, Adelaide
  - Trialworks Clinical Research Services, Brisbane
  - Dr Doongs Surgery, Burwood
  - Holdsworth House Medical Practice, Darlinghurst
  - Doctors of Ivanhoe,, Melbourne
  - Lung Institute of Western Australia,, Nedlands
  - Pitt Street Merrylands Medical Centre, Sydney
- New Zealand (7):
  - St George's Hospital, Christchurch, Christchurch
  - Bairds Road Family Health Care, Rotorua, Rotorua
  - Greenhithe Medical Centre, Auckland
  - Southern Clinical Trials Ltd, Christchurch
  - Caversham Medical Centre, Dunedin
  - Dr. Gillies, Rotorua
  - Hinemoa House Family Health Centre, Rotorua
- South Africa (34):
  - Jsha Research, Bloemfontein, Bloemfontein
  - Nortje, MD, Goodwood, Capetown
  - Greenbury Medical Centre, Greenbury, Durban
  - Sebastian, MD, Silverglen, Durban
  - Quinta-Research, Bloemfontein, Free State
  - Wilhase, AC, Reigerpark, Gauteg
  - NHC Medical Centre, Bryanston, Gauteng
  - R. Dulabh, MD, Klipspruit West, Gauteng
  - DJW Navorsing, Noordheuwel, Krugersdorp
  - Pillay, MD, Verulam, KwaZulu-Natal
  - Vawda, Z.FA, Durban, KZ-Natal
  - le Clus, MD, Kempton Park, Pretoria
  - Sunnyside Medi-Clinic, Sunnyside Pretoria, Pretoria
  - Kaapzicht Centre, Cape Town, W. Cape
  - Syzygy SMO Intercare Medical and Dental Centre, Cape Town, W. Cape
  - Clinical Project Research SA (Pty) Ltd., Worcester, W. Cape
  - Benmed Park Clinic, Benoni
  - Armansis Medical Centre, Brits
  - Cape Clinical Trial, Bishop Lavis Day Hospital, Cape Town
  - First House, Cape Town
  - Synapta Clinical Research Centre, Durban
  - Dr. Janari, Durban
  - Dr. van Rensburg, eManzimtoti
  - Dr. Makan, Johannesburg
  - Newgate Centre, Johannesburg
  - GCT Trials, Mercantile Hospital no 9, Port Elizabeth
  - Dr. Nel, Pretoria
  - Emmed Research, Pretoria
  - Dr. de Bruin, Pretoria
  - Westmed Clinical Trial Centre, Pretoria West Medicross Building, Pretoria
  - Dr. Fouche, Roodepoort
  - Dr. de Villiers, Scottburgh
  - Dr. Bhorat, Soweto
  - Clinical Projects Research SA Ltd, Worcester

RESULTS

PARTICIPANT FLOW:
Groups:
- Peramivir 600 mg: Peramivir 600 mg administered as bilateral 2-mL intramuscular injection.
Period: Overall Study
Arm/Group | Placebo | Peramivir 600 mg
Started | 203 | 202
Completed | 199 | 197
Not Completed | 4 | 5
Not completed — Lost to Follow-up | 3 | 3
Not completed — Did not receive study drug | 1 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT)
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Peramivir 600 mg | Total
Number analyzed (Participants) | 203 | 202 | 405
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (11.3) | 35 (12.1) | 35 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 102 | 206
  Male | 99 | 100 | 199
Race/Ethnicity, Customized [Number; unit: participants] — Participants may have been counted in more than 1 category; therefore, numbers may add up to more than the total number of participants.
  participants
    White or Caucasian | 101 | 106 | 207
    Black or African American | 68 | 61 | 129
    Asian | 15 | 15 | 30
    American Indian or Alaska Native | 5 | 3 | 8
    Other | 14 | 17 | 31
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.5 (6.73) | 27.2 (6.12) | 27.4 (6.43)
Estimated Time of Onset of Symptoms at Screening [Number; unit: participants]
  0-12 h Ago | 13 | 16 | 29
  12-24 h Ago | 91 | 81 | 172
  24-36 h Ago | 99 | 104 | 203
  Data Missing | 0 | 1 | 1
Initial Composite Symptom Score [Mean (Standard Deviation); unit: units on a scale] — Initial Composite Symptom Score is defined as the sum of the 7 symptoms of influenza initially recorded by the subject in the diary (cough; sore throat; nasal congestion; myalgia [aches and pains]; headache; feverishness; and fatigue), each graded on a 4-point severity scale [0, absent; 1, mild; 2, moderate; 3, severe]); for the composite score, individual scores were summed, with a range from 0 to 21.
  units on a scale | 14 (4.3) | 14 (3.9) | 14 (4.1)
Rapid Antigen Test (RAT) Results [Number; unit: participants] — Positive influenza infection confirmed by PCR or virus culture.
  participants
    Positive | 202 | 200 | 402
    No data reported | 1 | 2 | 3
Confirmed Influenza Infection Result [Number; unit: participants]
  Positive by PCR Only | 27 | 38 | 65
  Positive by Viral Culture Only | 0 | 0 | 0
  Positive by PCR and Viral Culture | 147 | 122 | 269
  Negative by PCR and Viral Culture | 28 | 40 | 68
  No Result/Sample | 1 | 2 | 3
Current Smoking Behavior [Number; unit: participants]
  Smoker | 37 | 37 | 74
  Nonsmoker | 166 | 165 | 331

OUTCOME MEASURES:

1. Primary Outcome: Time to Alleviation of Symptoms (Kaplan-Meier Estimate)
Description: The primary efficacy endpoint was the time to alleviation of symptoms calculated as the number of hours from initiation of study drug until the start of the time period in which all 7 symptoms of influenza were either absent or present at a level no greater than mild for at least 21.5 (24 hours - 10%) hours. Subjects with missing diary data were excluded and those who did not experience alleviation of symptoms were censored at the last observed symptom assessment.
Time Frame: Information collected twice daily beginning predose on Day 1 and through Day 9, then once daily through Day 14
Population: The Intent-to-Treat Infected with Influenza A (ITTI-A) population included all subjects who were randomized, received study drug, and had confirmed influenza A by culture or PCR.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Placebo | Peramivir 600 mg
Number analyzed (Participants) | 147 | 132
hours | 106.9 [90.4 to 127.4] | 91.1 [77.7 to 109.7]
Statistical Analysis 1: Comparison: Placebo vs Peramivir 600 mg; Test type: Superiority or Other; p = 0.222, Wilcoxon-Gehan test statistic; P-value is from a Wilcoxon-Gehan test statistic controlling for smoking status and hemisphere of enrollment; Hazard Ratio (HR) = 0.927, 95% CI 2-sided [0.723 to 1.188] — Hazard Ratio and corresponding 95% CI are based the Cox Regression Model including parameters for treatment, controlling for smoking status and hemisphere of enrollment

2. Secondary Outcome: Change in Influenza Virus Shedding
Description: Changes from Baseline in log10 TCID50/mL through Days 3, 4, and 9 were presented by treatment group for subjects with positive viral titers at Baseline (log10 TCID50/mL >0.5).
Time Frame: Baseline and Days 3, 4, 9
Population: The Intent-to-Treat Infected Influenza A (ITTI-A) population included all subjects who were randomized, received study drug, and had confirmed influenza A infection by culture or PCR.
Measure: Median (95% Confidence Interval); unit: log10(TCID50/mL)
Arm/Group | Placebo | Peramivir 600 mg
Number analyzed (Participants) | 120 | 97
log10(TCID50/mL)
  Change at Day 3 | -2.00 [-2.25 to -1.50] | -2.00 [-2.25 to -1.50]
  Change at Day 4 | -2.25 [-2.75 to -2.00] | -2.25 [-2.75 to -2.00]
  Change at Day 9 | -2.75 [-3.00 to -2.25] | -2.50 [-2.75 to -2.00]
Statistical Analysis 1: Comparison: Placebo vs Peramivir 600 mg; Test type: Superiority or Other; p > 0.05, van Elteren test; P-value for comparisons at all time points. P-value was based on the van Elteren test controlling for smoking status and hemisphere of enrollment

3. Other Pre Specified Outcome: Subject's Severity of Illness (Score*Hours)
Description: A subject's severity of illness (area under the symptom score curve, as measured in score-hours) was assessed using available symptom score data until the time of alleviation of symptoms.The score-hours were calculated as the product of the daily symptom score times the hours to alleviation. All available data until time of alleviation were utilized.
  The daily symptom score was defined as the sum of the 7 symptoms of influenza recorded by the subject in the diary each day (cough; sore throat; nasal congestion; myalgia [aches and pains]; headache; feverishness; and fatigue), each graded on a 4-point severity scale [0, absent; 1, mild; 2, moderate; 3, severe]); for the composite score, individual scores were summed, with a range from 0 to 21.
Time Frame: Information collected predose on Day 1 and then once daily through Day 14
Population: as for outcome 2
Measure: Median (Full Range); unit: score*hours
Arm/Group | Placebo | Peramivir 600 mg
Number analyzed (Participants) | 147 | 132
score*hours | 777.0 [18.0 to 3542.9] | 713.9 [23.5 to 4565.5]
Statistical Analysis 1: Comparison: Placebo vs Peramivir 600 mg; Test type: Superiority or Other; p = 0.421, van Elteren test; P-value is based on van Elteren test controlling for smoking status and hemisphere of enrollment

4. Other Pre Specified Outcome: Time to Resolution of Fever
Description: Time to resolution of fever was defined as the number of hours from initiation of study drug until temperature was less than 37.2 °C (99.0 °F) and no antipyretic medication had been taken for at least 12 hours.
Time Frame: Information collected twice daily beginning predose on Day 1 and through Day 9, then once daily through Day 14
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Placebo | Peramivir 600 mg
Number analyzed (Participants) | 147 | 132
hours | 44.7 [41.5 to 52.2] | 44.3 [40.1 to 55.5]
Statistical Analysis 1: Comparison: Placebo vs Peramivir 600 mg; Test type: Superiority or Other; p = 0.885, Wilcoxon-Gehan test statistic; P-values are from a Wilcoxon-Gehan test statistic controlling for smoking status and hemisphere of enrollment

5. Other Pre Specified Outcome: Incidence of Influenza-related Complications
Description: Study personnel were provided with an IRC checklist in the CRF to evaluate the subject for the presence of clinical signs and/or symptoms of the following IRCs: sinusitis, otitis, bronchitis, and pneumonia. Subjects with clinical signs and/or symptoms consistent with these conditions at Screening were not eligible for enrollment in this study.
Time Frame: 14 days
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | Peramivir 600 mg
Number analyzed (Participants) | 149 | 133
participants
  Any Influenza-Related Complication | 25 | 29
  Otitis | 2 | 4
  Sinusitis | 17 | 13
  Bronchitis | 10 | 15
  Pneumonia | 0 | 3
Statistical Analysis 1: Comparison: Placebo vs Peramivir 600 mg; Test type: Superiority or Other; p = 0.306, Cochran-Mantel-Haenszel; P-value is based on the Cochran-Mantel-Haenszel general association test controlling for smoking status and hemisphere of enrollment

6. Other Pre Specified Outcome: Baseline Influenza Virus A (H1N1) Susceptibility to Neuraminidase Inhibitors (Mean IC50)
Description: Baseline value of influenza virus susceptibility to neuraminidase inhibitors was assessed using virology laboratory tests. Virology laboratory tests included phenotypic characterizations of influenza virus recovered (hemagglutinin and neuraminidase) and viral susceptibility to zanamivir, oseltamivir, and peramivir, as well as genotyping of virus isolates.
Time Frame: Baseline
Population: A subgroup of the Intent-to-Treat Infected Influenza A (ITTI-A) population that included all subjects who were randomized, received study drug, and had confirmed influenza A (H1N1) infection by culture or PCR. N was 113 for zanamivir susceptibility in the Placebo group.
Measure: Mean (Standard Error); unit: nM
Arm/Group | Placebo | Peramivir 600 mg
Number analyzed (Participants) | 114 | 89
nM
  A: H1N1-Baseline Peramivir Susceptibility | 67.46 (54.625) | 72.27 (88.306)
  A: H1N1-Baseline Oseltamivir Susceptibility | 983.41 (1129.29) | 1007.29 (1425.095)
  A: H1N1-Baseline Zanamivir Susceptibility | 1.27 (1.131) | 1.48 (1.686)

7. Other Pre Specified Outcome: Change in Influenza Virus A (H1N1) Susceptibility to Neuraminidase Inhibitors (Fold Change From Baseline in IC50)
Description: Change from Baseline to last positive value of influenza virus susceptibility to neuraminidase inhibitors was assessed using virology laboratory tests. Virology laboratory tests included phenotypic characterizations of influenza virus recovered (hemagglutinin and neuraminidase) and viral susceptibility to zanamivir, oseltamivir, and peramivir, as well as genotyping of virus isolates. These analyses were presented separately by treatment group and viral subtype.
Time Frame: Baseline and up to 14 days
Population: A subgroup of the Intent-to-Treat Infected Influenza A (ITTI-A) population that included all subjects who were randomized, received study drug, and had confirmed influenza A (H1N1) infection by culture or PCR. N is for fold change (participants who had baseline and last positive susceptibility values to zanamivir, oseltamivir, and peramivir).
Measure: Mean (Standard Error); unit: Fold Change from Baseline
Arm/Group | Placebo | Peramivir 600 mg
Number analyzed (Participants) | 39 | 37
Fold Change from Baseline
  A: H1N1- Fold Change in Peramivir Susceptibility | 1.03 (0.660) | 1.10 (0.677)
  A: H1N1- Fold Change in Oseltamivir Susceptibility | 1.20 (1.055) | 1.28 (1.441)
  A: H1N1- Fold Change in Zanamivir Susceptibility | 3.68 (11.882) | 2.67 (9.797)

8. Other Pre Specified Outcome: Baseline Influenza Virus B Susceptibility to Neuraminidase Inhibitors (Mean Baseline IC50)
Description: Baseline value of influenza virus susceptibility to neuraminidase inhibitors was assessed using virology laboratory tests. Virology laboratory tests included phenotypic characterizations of influenza virus recovered (hemagglutinin and neuraminidase) and viral susceptibility to zanamivir, oseltamivir, and peramivir, as well as genotyping of virus isolates. Baseline was defined as the last non-missing value occuring prior to the initiation of study drug.
Time Frame: Baseline and up to 14 days
Population: A subgroup of the Intent-to-Treat Infected (ITTI) population that included all subjects who were randomized, received study drug, and had confirmed influenza B infection by culture or PCR. The n reported is the number of participants who had baseline susceptibility values to zanamivir, oseltamivir, and peramivir.
Measure: Mean (Standard Error); unit: nM
Arm/Group | Placebo | Peramivir 600 mg
Number analyzed (Participants) | 23 | 24
nM
  B: Baseline Peramivir Susceptibility | 6.47 (2.442) | 6.03 (3.633)
  B: Baseline Oseltamivir Susceptibility | 40.98 (24.202) | 28.72 (17.838)
  B: Baseline Zanamivir Susceptibility | 5.78 (2.682) | 4.65 (2.282)

9. Other Pre Specified Outcome: Change in Influenza Virus B Susceptibility to Neuraminidase Inhibitors (Mean Baseline IC50 and Fold Change From Baseline in IC50)
Description: Change from Baseline to last positive value of influenza virus susceptibility to neuraminidase inhibitors was assessed using virology laboratory tests. Virology laboratory tests included phenotypic characterizations of influenza virus recovered (hemagglutinin and neuraminidase) and viral susceptibility to zanamivir, oseltamivir, and peramivir, as well as genotyping of virus isolates. These analyses were presented separately by treatment group and viral subtype. Baseline was defined as the last non-missing value occuring prior to the initiation of study drug.
Time Frame: Baseline and up to 14 days
Population: A subgroup of the Intent-to-Treat Infected (ITTI) population that included all subjects who were randomized, received study drug, and had confirmed influenza B infection by culture or PCR. The n reported is the number for fold change (participants who had baseline and last positive susceptibility values to zanamivir, oseltamivir, and peramivir).
Measure: Mean (Standard Error); unit: Fold Change from Baseline
Arm/Group | Placebo | Peramivir 600 mg
Number analyzed (Participants) | 8 | 12
Fold Change from Baseline
  B: Fold Change in Peramivir Susceptibility | 1.27 (1.319) | 0.92 (0.442)
  B: Fold Change in Oseltamivir Susceptibility | 1.24 (0.819) | 0.95 (0.374)
  B: Fold Change in Zanamivir Susceptibility | 1.10 (0.737) | 0.95 (0.497)

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs included any AEs that occurred after treatment on Day 1 and up to and including the visit on Day 14.
Description: Three of 405 subjects were randomized but did not receive treatment and were therefore not included in the safety population (N = 402; 202 in the Placebo group and 200 in the Peramivir 600 mg group).
Arm/Group | Placebo | Peramivir 600 mg
Serious Adverse Events (participants affected / at risk) | 1/202 | 0/200
Other Adverse Events (participants affected / at risk) | 27/202 | 31/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=202) | Peramivir 600 mg (N=200)
Disseminated Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=202) | Peramivir 600 mg (N=200)
Nausea (Gastrointestinal disorders) | 10 | 7
Diarrhoea (Gastrointestinal disorders) | 8 | 6
Vomiting (Gastrointestinal disorders) | 0 | 4
Blood creatine phosphokinase increased (Investigations) | 1 | 11
Injection site pain (General disorders) | 2 | 4
Urinary tract infection (Infections and infestations) | 5 | 1
Headache (Nervous system disorders) | 5 | 0

LIMITATIONS AND CAVEATS:
The majority of the subjects enrolled in this study with a laboratory confirmed influenza infection were infected with an influenza A/H1N1 virus containing an H275Y mutation associated with reduced susecptibility to peramivir and oseltamivir.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No